CLINICAL TRIAL: NCT03911271
Title: Low-dose Atropine for the Prevention of Myopia Progression in Danish Children - a Randomized, Double-masked, Multicenter, 36-month Prospective 1:1:1 Study of Safety and Efficacy of 0.1% Atropine Loading Dose to Single 0.01% Atropine and Placebo
Brief Title: Low-dose Atropine for the Prevention of Myopia Progression in Danish Children
Acronym: APP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Line Kessel (Other)
Collaborators: Aarhus University Hospital (Other); Vejle Hospital (Other)
Responsible Party: Sponsor-Investigator, Line Kessel, Consultant ophthalmologist, Associate Professor, MD, Ph.D., FEBO, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Line Kessel, RH-Glostrup
Record Dates: First submitted 2019-04-02; First posted 2019-04-11 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine; Contraceptives, Oral; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Loading dose (Experimental): In phase 1 (treatment phase), the participants (n=33) will receive 0.1% atropine loading dose for 6 months followed by 0.01 % atropine for 18 months. The eye drops are administered as one eye drop daily in each eye at bedtime.
  In phase 2 (washout phase), treatment will be stopped and the participants monitored for 12 months.
  Interventions: Drug: 0.1% atropine and 0.01% atropine
- Low dose (Experimental): In phase 1 (treatment phase), the participants (n=32) will receive 0.01 % atropine for 24 months. The eye drops are administered as one eye drop daily in each eye at bedtime.
  In phase 2 (washout phase), treatment will be stopped and the participants monitored for 12 months.
  Interventions: Drug: 0.01% atropine
- Placebo (Placebo Comparator): In phase 1 (treatment phase), the participants (n=32) will receive placebo eye drops for 24 months. The eye drops are administered as one eye drop daily in each eye at bedtime.
  In phase 2 (washout phase), treatment will be stopped and the participants monitored for 12 months.
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: 0.1% atropine and 0.01% atropine — 0.1% atropine loading dose for 6 months followed by 0.01% atropine for 18 months
  Other Names: Loading dose
  Arms: Loading dose
Drug: 0.01% atropine — 0.01% atropine for 24 months
  Other Names: Low-dose
  Arms: Low dose
Drug: 0.9% Sodium-chloride — Placebo for 24 months
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Myopia (nearsightedness) is increasing in prevalence throughout the world. It is associated with a risk of potentially blinding complications such as retinal detachment and myopic maculopathy. There is a direct association between the degree of myopia and the risk of complications. Myopia develops in childhood and during adolescence. To prevent higher degrees of myopia, we need to halt disease progression in children and teenagers. Low-dose atropine eye drops have been shown to reduce myopia progression by 50% in Asian populations but its effect in non-Asian populations is unknown. The aim of this study is to investigate if low-dose atropine can reduce myopia progression in Danish children and teenagers. The study is an investigator initiated randomized clinical trial conducted as a collaboration between three Danish Eye Departments covering all of Denmark.

DETAILED DESCRIPTION:
The main hypotheses tested in this study are:

* 0.01% atropine one drop nightly reduces the progression of childhood myopia in Danish children.
* 0.01% atropine one drop nightly is safe and with no significant side effects.
* A 6-month loading dose of 0.1% atropine followed by a 0.01% atropine maintenance dose is superior to single 0.01% atropine.
* 0.1% atropine one drop nightly is safe and has tolerable side effects.
* The rebound effect after stopping both atropine regimens is limited.
* Choroidal thickness is a predictor for the progression of childhood myopia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged ≥6-<9 years: myopia ≤-1 (spherical power) in at least one eye
* Children aged ≥9-≤12 years: myopia ≤-2 (spherical power) in at least one eye
* Cylinder less than 1.5 diopters

Exclusion Criteria:

* Myopia related to retinal dystrophies
* Collagen syndroms (Ehlers-Danlos syndrome, Marfan syndrome and Stickler syndrome)
* Other ocular pathology (e.g., amblyopia, strabismus)
* Previous eye surgery
* Previous use of agents thought to affect myopia progression, e.g. atropine, pirenzepine or 7-methylxanthine (metabolite of caffeine and theobromine) and orthokeratology contact lenses
* Known allergy to atropine or any of the contents of the trial medication (active and in-active ingredients) used in the study
* Non-compliance to eye examinations
* Serious systemic health troubles (e.g., cardiac or respiratory illness) and developmental disorders and delays

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Department of Ophthalmology, Aarhus University Hospital, Aarhus
  - Department of Ophthalmology, Rigshospitalet-Glostrup, Glostrup Municipality
  - Department of Ophthalmology, Vejle Hospital, Vejle

REFERENCES:
- [Derived] Hansen NC, Hvid-Hansen A, Bek T, Moller F, Jacobsen N, Kessel L. The Macular Choroidal Thickness in Danish Children with Myopia After Two-Year Low-Dose Atropine and One-Year Wash-Out: A Placebo-Controlled, Randomized Clinical Trial. Ophthalmol Ther. 2024 Dec;13(12):3111-3122. doi: 10.1007/s40123-024-01051-5. Epub 2024 Oct 18. PMID 39422837
- [Derived] Hansen NC, Hvid-Hansen A, Moller F, Bek T, Larsen DA, Jacobsen N, Kessel L. Safety and efficacy of 0.01% and 0.1% low-dose atropine eye drop regimens for reduction of myopia progression in Danish children: a randomized clinical trial examining one-year effect and safety. BMC Ophthalmol. 2023 Oct 30;23(1):438. doi: 10.1186/s12886-023-03177-9. PMID 37904082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Danish children with myopia were referred from optometrists and ophthalmologists across Denmark.
  Recruitment and follow-up took place between May 2019 and April 2024 (Last patient last visit = 23 of April 2024)
Period: Overall Study
Arm/Group | Loading Dose | Low Dose | Placebo
Started | 33 | 32 | 32
Completed | 31 | 31 | 29
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data is reported per arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Loading Dose | Low Dose | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 32 | 97
Age, Continuous [Mean (Full Range); unit: Years] — Mean Age per Group and Full Range
  Years | 9.5 [6 to 12] | 9.4 [7 to 12] | 9.2 [6 to 12] | 9.4 [6 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 18 | 55
  Male | 14 | 14 | 14 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 32 | 32 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Axial length [Mean (Standard Deviation); unit: mm] — Means are reported per arm
  mm | 24.5 (0.86) | 24.6 (0.78) | 24.4 (0.90) | 24.6 (0.84)
Spherical equivalent refraction [Mean (Standard Deviation); unit: Diopters] — Means are reported per arm
  Diopters | -3.00 (1.59) | -2.97 (1.13) | -3.07 (1.04) | -2.99 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Axial Length at 36 Months
Description: Treatment group comparison of axial length at 36 months, as measured using IOLMaster 700
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Loading Dose: In phase 1 (treatment phase), the participants (n=50) will receive 0.1% atropine loading dose for 6 months followed by 0.01 % atropine for 18 months. The eye drops are administered as one eye drop daily in each eye at bedtime.
  In phase 2 (washout phase), treatment will be stopped and the participants monitored for 12 months.
- Low Dose: In phase 1 (treatment phase), the participants (n=50) will receive 0.01 % atropine for 24 months. The eye drops are administered as one eye drop daily in each eye at bedtime.
  In phase 2 (washout phase), treatment will be stopped and the participants monitored for 12 months.
- Placebo: In phase 1 (treatment phase), the participants (n=50) will receive placebo eye drops for 24 months. The eye drops are administered as one eye drop daily in each eye at bedtime.
  In phase 2 (washout phase), treatment will be stopped and the participants monitored for 12 months.
Arm/Group | Loading Dose | Low Dose | Placebo
Number analyzed (Participants) | 31 | 31 | 29
mm | 25.28 [25.06 to 25.50] | 25.25 [25.03 to 25.47] | 25.33 [25.11 to 25.56]

2. Primary Outcome: Spherical Equivalent at 36 Months
Description: Treatment group comparison of spherical equivalent at 36 months, as measured using cycloplegic autorefraction
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: Diopters
Arm/Group | Loading Dose | Low Dose | Placebo
Number analyzed (Participants) | 31 | 31 | 29
Diopters | -4.45 [-4.84 to -4.06] | -4.26 [-4.65 to -3.87] | -4.43 [-4.83 to -4.03]

3. Secondary Outcome: Adverse Events
Description: Total individual adverse events per interventional arm
Time Frame: 36 months
Measure: Number; unit: Number of adverse events reported
Arm/Group | Loading Dose | Low Dose | Placebo
Number analyzed (Participants) | 33 | 32 | 32
Number of adverse events reported | 104 | 22 | 18

4. Secondary Outcome: Change in Choroidal Thickness From Baseline to 36 Months
Description: Treatment group comparison of change in choroidal thickness from baseline to 36 months, as measured using optical coherence tomography (OCT)
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Loading Dose | Low Dose | Placebo
Number analyzed (Participants) | 33 | 32 | 32
microns | 2 [-11 to 15] | 7 [-3 to 17] | 3 [-8 to 14]

ADVERSE EVENTS:
Time Frame: From enrollment to three years
Description: The intent is to report the total number of adverse events AND reactions.
  Adverse events and reactions that are considered normal reactions to an eye examination (including stinging when applying eye drops for the examinations and short-term photophobia and blurred vision following eye examination) was not considered an AE/AR.
  Examples of adverse events that are exempted from registration includes conditions that are common to normal child development and child life were not reported.
Arm/Group | Loading Dose | Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32 | 3/32
Other Adverse Events (participants affected / at risk) | 33/33 | 10/32 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loading Dose (N=33) | Low Dose (N=32) | Placebo (N=32)
Lymphadenopathy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Deemed not related to the study drug
Suspicion of meningitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Suspicion was later abated
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Deemed not related to the study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loading Dose (N=33) | Low Dose (N=32) | Placebo (N=32)
Eye redness/irritation (Eye disorders) | 8 (8) | 6 (6) | 5 (5)
Photophobia (Eye disorders) | 30 (30) | 4 (4) | 1 (1)
Other (Eye disorders) | 14 (14) | 10 (10) | 11 (11)
Blurred near vision (Eye disorders) | 33 (33) | 2 (2) | 1 (1) — Participants were asked whether they experienced near vision blur
Blurred distance vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) — Participants were asked whether they experienced distance vision blur
Dilated pupils (Eye disorders) | 19 (19) | 0 (0) | 0 (0) — Participants were asked whether they experienced dilated pupils

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03911271/Prot_SAP_000.pdf